CLINICAL TRIAL: NCT04662671
Title: Phase I/II Randomized, Dose Escalation Study to Evaluate the Safety and Antiviral Activity of the RD-X19 Device in SARS-CoV-2 Infected Individuals With Uncomplicated COVID-19
Brief Title: Phase I/II Safety, Dose Finding & Antiviral Activity of RD-X19 in Mild/Moderate Outpatient COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmitBio Inc. (Industry)
Responsible Party: Sponsor
Organization: KNOWBio Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB-P12-01
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a randomized, double-blind, sham-controlled study in SARS-CoV-2 infected individuals with outpatient COVID-19. Subjects will be randomized 2:1 RD-X19 to Sham Device treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RD-X19 Device (Experimental): Experimental device that uses safe electromagnetic energy to stimulate the proximal repository of respiratory tract infectious disease pathogens.
  Interventions: Device: RD-X19
- Sham Device (Sham Comparator): Investigational device that uses safe electromagnetic energy to target the oropharynx but at energy levels with a lower inactivation potential against SARS-CoV-2 in vitro.
  Interventions: Device: RD-X19

INTERVENTIONS:
Device: RD-X19 — Experimental device that uses safe electromagnetic energy to stimulate the proximal repository of respiratory tract infectious disease pathogens.

SUMMARY:
This randomized, Phase I/II feasibility study will evaluate the safety and efficacy of the RD-X19 device in SARS-CoV-2 infected individuals with uncomplicated COVID-19.

DETAILED DESCRIPTION:
This is a randomized, sham-controlled dose escalation and bioeffect study. The primary goal of the study is to evaluate the safety of the RD-X19 device in SARS-CoV-2 infected individuals with outpatient COVID-19 and to assess the reduction of SARS-CoV-2 viral load in each dose group compared to sham controls.

The primary safety measure is absence of device-related serious adverse events or patterns of severity ≥2 device-related adverse events. Safety and tolerability (local reactogenicity) will be assessed actively on each clinic visit by review of potential adverse events (AEs) and targeted physical examination, as required. Metabolic, liver, kidney and hematological laboratory evaluations will be performed at baseline and at Day 8 or early termination (and potentially during unscheduled) clinic visits.

Methemoglobin assessments will be performed at baseline and Day 8.

Various efficacy assessments will explore the impact of RD-X19 treatment on the reduction in log10 SARS-CoV-2 viral load and alleviation of symptoms associated with COVID-19. Both the magnitude of reduction as a function of dose as well as time to clearance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for SARS-CoV-2 antigen via nasal swab at or within the past 24 hours of the screening visit detected using an FDA authorized SARS-CoV-2 antigen test.
2. Onset of signs and symptoms consistent with COVID-19* no longer than within the past 3 days* and have either a) a fever of at least 100 °F or b) at least two moderate or severe symptoms (cough, sore throat, nasal congestion, headache, chills/sweats, muscle or joint pain, fatigue, and nausea) at the time of screening.
3. Provides written informed consent prior to initiation of any study procedures.
4. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
5. Agrees to the collection of nasopharyngeal swabs, oropharyngeal swabs, oral saliva specimen collection and venous blood specimens per protocol.
6. Agrees to refrain from using oral antiseptics (e.g. hydrogen peroxide rinse, Listerine) or mouthwashes of any kind during the study.
7. Male or non-pregnant female, 18 to 65 years of age, inclusive, at time of enrollment.
8. No uncontrolled disease process (chronic or acute), other than COVID-19 signs and symptoms*.
9. No physical or mental conditions or attributes at the time of screening, which in the opinion of the PI, will prevent full adherence to, and completion of, the protocol.

Exclusion Criteria:

1. Positive urine pregnancy test at screening.
2. Any medical disease or condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.
3. Presence of self-reported or medically documented uncontrolled significant medical or psychiatric condition(s) other than COVID-19.
4. Reports a recent positive test result (within the past 6 months) for hepatitis B surface antigen, hepatitis C virus antibody, or HIV-1 antibodies at screening.
5. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 1 month of Study Day 1.
6. COVID-19 signs associated with acute respiratory distress or imminent serious medical outcomes. ^^
7. BMI ≥36
8. Subjects living (e.g., siblings, spouses, relatives, roommates) in the same household cannot be enrolled.
9. Has participated in another investigational study involving any intervention for SARS-CoV-2/COVID- 19 within the past 6 months or any clinical trial with interventional investigational product within 30 days of screening.
10. Currently enrolled in or plans to participate in another clinical trial with an interventional investigational agent that will be received during the studyperiod.
11. History of hospitalization within the past 60 days.
12. History of systemic antiviral therapies within the past 30 days.
13. History of oral corticoid steroid use within the past 14 days or steroid injection within the past 6 months. Active use of nasal or inhalable steroids is also exclusionary. Topical steroids are not exclusionary.
14. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to nitrites, nitrates, or sun exposure.
15. Has any oral abnormality (e.g. ulcer, oral mucositis, gingivitis) that in the opinion of the investigator would interfere with device use, or intra-oral metal body piercings that cannot be removed for the duration of the study. Metal orthodontia is permitted as braces will be covered by the device mouthpiece.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EB-P12-01 Study Director, Study Director — EmitBio
Locations (2):
- United States (2):
  - Site 2, Miami, Florida
  - Site 1, College Station, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: Sham: The sham devices were designed to provide the same user experience but at energy and fluence levels with a lower inactivation potential against SARS-CoV-2 in vitro than that delivered by the active devices.
Period: Overall Study
Arm/Group | RD-X19 Device | Sham
Started | 20 | 11
Completed | 20 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RD-X19 Device | Sham | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 11 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnic Group: Hispanic or Latino | 15 | 7 | 22
  Race or Ethnic Group: White | 4 | 3 | 7
  Race or Ethnic Group: Black | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 11 | 31
Laboratory Confirmed SARS-CoV-2 at Baseline via RT-PCR (saliva) [Count of Participants; unit: Participants] | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Measure
Description: Number of Participants with device-related serious adverse events or any patterns of severity ≥2 device-related adverse events in the same SOC grouping of Preferred Terms based on Medical Dictionary for Regulatory Activities (MedDRA) coding, as determined throughout the course of the study.
Time Frame: Baseline thru Day 8
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device | Sham
Number analyzed (Participants) | 20 | 11
Participants | 0 | 0

2. Primary Outcome: Primary Efficacy Measure
Description: Time weighted average change in viral load from baseline by RT-qPCR from Day 1 to Day 8.
Time Frame: Baseline to Day 8
Population: Modified Analysis Set with Laboratory Confirmed SARS-CoV-2 at Baseline via RT-PCR
Measure: Least Squares Mean (95% Confidence Interval); unit: TWAC (SARS-COV-2 N1 Log10 copies/mL)
Arm/Group | RD-X19 Device | Sham
Number analyzed (Participants) | 17 | 11
TWAC (SARS-COV-2 N1 Log10 copies/mL) | -1.69 [-2.27 to -1.12] | -1.23 [-1.95 to -0.52]

3. Secondary Outcome: Proportion of Subjects Demonstrating Clearance of Viral Infection
Description: Proportion of subjects demonstrating clearance of viral infection, defined as a negative test via RT-qPCR on Day 8/ET.
Time Frame: Days 1, 3, 5 and 8
Population: Modified analysis set for virologic efficacy assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device | Sham Device
Number analyzed (Participants) | 17 | 11
Participants | 10 | 4

4. Secondary Outcome: Median Time to Alleviation of Symptoms
Description: Median time to alleviation of symptoms as measured by the time when all eight symptoms (cough, sore throat, nasal congestion, headache, chills/sweats, muscle or joint pain, fatigue, and nausea) had been assessed by the subject as none (0) or mild (1).
Time Frame: Daily through day 8
Population: ITT
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | RD-X19 Device | Sham
Number analyzed (Participants) | 20 | 11
hours | 75.3 [48.3 to 117.2] | 112.7 [38.0 to 166.2]

5. Post Hoc Outcome: Median Time to Sustained Resolution of Symptoms
Description: Median time to Sustained Resolution of Symptoms as measured by the time when all eight symptoms (cough, sore throat, nasal congestion, headache, chills/sweats, muscle or joint pain, fatigue, and nausea) had been assessed by the subject as none (0) or mild (1) without rebound of any score greater than 1 for the remainder of the trial.
Time Frame: Daily through day 8
Population: ITT
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | RD-X19 Device | Sham
Number analyzed (Participants) | 20 | 11
hours | 103.8 [69.0 to 130.8] | 160.7 [38.0 to 192]

ADVERSE EVENTS:
Time Frame: 8 Days
Arm/Group | RD-X19 Device | Sham
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 12/20 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD-X19 Device (N=20) | Sham (N=11)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Chills (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by signed Non-confidentiality Agreements and Clinical Trial Agreements with EmitBio, Inc. as the sponsor of this trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT04662671/Prot_SAP_000.pdf